CLINICAL TRIAL: NCT01599013
Title: Randomized Phase II Study Assessing the Combination of Vinflunine With Gemcitabine and Vinflunine With Carboplatin in Patients Ineligible to Cisplatin With Advanced or Metastatic Transitional Cell Carcinoma of the Urothelium
Brief Title: JAVLOR Association Study in CDDP-unfit Patients With Advanced Transitional Cell Carcinoma: Gemcitabine Versus Carboplatin
Acronym: JASINT1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L00070 IN 213 P1
Record Dates: First submitted 2012-04-16; First posted 2012-05-15 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Bladder Transitional Cell Carcinoma Stage IV
Keywords: urothelial carcinoma; bladder cancer; vinflunine; transitional cell carcinoma; advanced or metastatic; unfit; ineligible to cisplatin; renal impairment; renal insufficiency; urologic neoplasms; urogenital neoplasm; urinary neoplasms; cisplatin; tubulin inhibitors
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms; Neoplasm Metastasis; Renal Insufficiency; Urologic Neoplasms; Urogenital Neoplasms | interventions — vinflunine; Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vinflunine plus Gemcitabine (Other)
  Interventions: Drug: Vinflunine, Gemcitabine
- Vinflunine plus Carboplatin (Other)
  Interventions: Drug: Vinflunine, Carboplatin

INTERVENTIONS:
Drug: Vinflunine, Gemcitabine — * Vinflunine 280 or 250 mg/m2, IV administration over 20 minutes (starting dose based on baseline creatinine clearance value), Day 1 every 3 weeks up to progression or unacceptable toxicity or patient's refusal
  * Gemcitabine 750 or 1000 mg/m2, IV administration over 30 minutes (starting dose based on baseline creatinine clearance value), Day 1 and 8 every 3 weeks up to progression or unacceptable toxicity or patient's refusal
  Other Names: JAVLOR, GEMZAR
  Arms: Vinflunine plus Gemcitabine
Drug: Vinflunine, Carboplatin — * Vinflunine 280 or 250 mg/m2, IV administration over 20 minutes (starting dose based on baseline creatinine clearance value), Day 1 every 3 weeks up to progression or unacceptable toxicity or patient's refusal
  * Carboplatin AUC 4.5, IV administration over 60 minutes, Day 1 every 3 weeks up to progression or unacceptable toxicity or patient's refusal
  Other Names: JAVLOR, CBDCA
  Arms: Vinflunine plus Carboplatin

SUMMARY:
This study is assessing the combination of well known cytotoxics with a novel anti-cancer agent that could be administered as monotherapy without renal toxicity in patients with renal impairment presenting with advanced or metastatic urothelial carcinoma previously treated with a platinum-based regimen. The intent of this study is to clarify the benefit/risk ratio of the two most promising associations of cytotoxics including the novel therapeutic agent, vinflunine: vinflunine-gemcitabine and vinflunine-carboplatin.

DETAILED DESCRIPTION:
Gemcitabine and carboplatin have been the most studied and used anticancer agents in cisplatin-unfit patients with advanced urothelial carcinoma. Both agents previously demonstrated clinical activity as single agent and/or as part of combination regimen in patients with advanced or metastatic disease even if clinical benefits and survival remains limited in this setting for this population.

The purpose of this study is to test in a randomized trial enrolling patients with renal impairment or moderate congestive heart failure two combinations of a novel cytotoxic agent, vinflunine, one with gemcitabine and another with carboplatin in order to determine the most promising combination in the first line treatment of advanced/metastatic urothelial carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged ≥ 18 years and < 80 years
* Signed written informed consent
* Histologically confirmed diagnosis of locally advanced or metastatic predominantly transitional cell carcinoma of the urothelium (TCCU)
* Ineligibility for cisplatin-based therapy because of at least one of the following two medical conditions:

  * Calculated creatinine clearance (Cockcroft-Gault formula)< 60 mL/min
  * New York Heart Association Classification Stage II-III Congestive Heart Failure (documented by medical history)
* "Measurable" disease with at least one uni-dimensional lesion according to RECIST guideline (version 1.1)
* ECOG performance status of 0 or 1
* Estimated life expectancy of at least 12 weeks
* Patient without prior systemic anticancer therapy unless if it had been administered as neoadjuvant or adjuvant chemotherapy (CT) for TCCU and if the patient has documented relapse ≥ 6 months after the last dose of CT (prior intravesical CT allowed)
* Adequate bone marrow and hepatic functions as evidenced by:

  * Absolute Neutrophil Count ≥ 2,000/mm3 (≥ 2.0 x 109/L)
  * Haemoglobin ≥ 10 g/dL
  * Platelet count ≥ 100,000/mm3
  * Serum total bilirubin ≤ 1.5 x upper limit of normal (ULN)
  * Transaminases ≤ 2.5 x ULN [≤ 5 x ULN only in case of liver metastasis]
* Absence of psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; these conditions should be assessed with the patient before registration in the trial

Exclusion Criteria:

* ECOG performance status ≥ 2
* Woman if pregnant or lactating or with positive pregnancy test at inclusion; woman of child-bearing potential who did not use or is unwilling or unable to use an acceptable method to avoid pregnancy during the 2 months preceding the start of study treatment, for the entire study period and for up to 3 months after the last dose of study treatment; sexually active fertile man not using effective birth control during the study and up to 6 months after the last dose of study treatment if his partner is a woman of child-bearing potential
* Known brain metastasis or leptomeningeal involvement.
* Peripheral neuropathy Grade ≥ 2 by NCI CTC
* Prior radiation to ≥ 30% of the bone marrow or completed < 30 days ago or without full recovery of toxicities
* Other serious illness or medical condition including:

  * Infection requiring systemic anti-infective therapy
  * Any medical condition that might not be controlled, for instance patients with unstable angina, patients with myocardial infarction within 6 months or uncontrolled diabetes
* Prior systemic chemotherapy for advanced or metastatic disease or neoadjuvant/adjuvant chemotherapy that was completed < 6 months before documented progression
* Patient who had received any other investigational drug or anti-cancer therapy within 30 days before randomisation
* Other malignancies except adequately treated basal carcinoma of the skin, in-situ cervix carcinoma, localised prostate cancer with limited risk of recurrence (pT ≤ 2b, Gleason score ≤ 7) that was incidentally discovered and did not lead to any other treatment apart from prostatectomy, or any other tumor with a disease free interval ≥ 5 years
* Inadequate renal function defined by a serum creatinine clearance < 30 mL/min (Cockcroft-Gault formula)
* Known hypersensitivity to the study drugs or to drugs with similar chemical structures
* Patients who require treatment with ketoconazole, itraconazole, ritonavir, amprenavir, indinavir, rifampicin (any potent CYP3A4 inhibitor or inducer) or phenytoin
* Any concurrent chronic system immune therapy or previous organ allograft
* Electrocardiogram (ECG) with significant modifications suggesting a high risk of occurrence of an acute clinical event

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2011-02; Primary Completion 2013-10 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Disease control rate as defined by RECIST criteria (version 1.1) as a percentage of best overall responses of Complete (CR) + Partial (PR) + Stable Disease (SD) for both Vinflunine-Gemcitabine and Vinflunine-Carboplatin combinations | Change from baseline in tumor assessment at 12 weeks (cycle 4)
  Assessment of lesions (measurable and non-measurable) should be performed at baseline and every 6 weeks (assessment interval).
  Evaluable patients: all baseline lesions must have been assessed at least once after the second cycle (6 weeks); patients who progress before the first evaluation will be considered as early progression.
  Primary analysis is planned on the intent to treat population, secondary analysis being performed on the evaluable population.

SECONDARY OUTCOMES:
Tumor Response Rate as defined by RECIST criteria (version 1.1) with a best response as Complete (CR) or Partial (PR) | Change from baseline in tumor assessment at 12 weeks (cycle 4)
  Assessment of lesions (measurable and non-measurable) should be performed at baseline and every 6 weeks (assessment interval).
  Evaluable patients: all baseline lesions must have been assessed at least once after the second cycle (6 weeks); patients who progress before the first evaluation will be considered as early progression.
Duration of Disease control in Participants With Best Response of CR + PR + SD | From the date of randomisation until the date of documented progression or date of death due to any cause, assessed up to 10 months
  Tumor assessment at baseline and then every 6 weeks, until tumor progression. Duration of disease control according to investigator will be calculated among the responders and stable patients from the date of randomisation until the documentation of progression or death due to any cause. Patients who are lost to follow-up without progression, or reach the time point of analysis without a known record of progression or death will have the duration of disease control censored at the date of last tumour assessment or last contact of a follow-up showing no progression, whichever occur last.
Duration of Response in Participants With Best Response of CR or PR | From the date that measurement criteria are first met for complete or partial response until the date of documented progression or date of death due to any cause, assessed up to 10 months
  Tumor assessment at baseline and then every 6 weeks, until tumor progression. Duration of response will be calculated among the responders (i.e. CR and PR) . Patients who are lost to follow-up, or reach the time point of analysis without a known record of progression or death will have the duration of response censored at the date of last tumour assessment or last contact of a follow-up showing no progression, whichever occur last.
Time to First Response calculated among the responders | From the date of randomisation up to the first report of documented response, assessed up to 12 weeks (cycle 4).
  Tumor assessment at baseline and then every 6 weeks. Will be calculated among the responders (i.e. CR and PR)
Time to Treatment Failure | From the date of randomisation until tumor progression, unacceptable toxicity, withdrawal of patient consent, lost to follow-up or start of new anticancer therapy, assessed up to 10 months.
  Tumor assessment (RECIST) every 6 weeks. Patients who reach the time point of analysis without failure as defined above will have the time to treatment failure censored at the date of last tumour assessment or last contact of a follow-up not showing progression. Patients who discontinued treatment for other reason and who are lost to follow-up will be censored at the date of last contact.
Progression Free Survival | From the date of randomisation until the date of progression or the date of death from any cause if no progression was recorded before, median patient follow-up of 11 months
  Tumor assessment every 6 weeks (RECIST).Patients who are lost to follow-up, or reach the time point of analysis without a known record of progression or death will have the progression-free survival censored at the date of last tumour assessment or last contact of a follow-up showing no progression, whichever occur last.
Overall Survival | From the time of randomisation up to death or last follow-up, assessed with a median patient follow-up of 15 months (assessed up to 24 months)
  Data recording every 3 months. For patients who have not died, survival time will be censored at the date of last news (i.e: date of last administration, tumor assessment, clinical examination, haematological or biochemistrical assessment or date of last contact).
Number of Participants With Serious Adverse Events (SAEs), Adverse Events (AEs) and AEs Leading to Discontinuation | AE and SAE will be collected up to 30 days after the last treatment administration, on an expected average period of 17 weeks
  Population: all treated patients unless the patient is lost to follow-up immediately after the start of the treatment. The patients will be analysed in the treatment arm they actually received.
  The NCI-CTC classification version 2.0 will be used to classify toxicities. Maximum grade or severity will be reported by cycle and by patient for each MedDRA Preferred Term. Analyses will be performed both regardless the relationship to treatment and related to treatment.
  Biochemical toxicities: the worst CTCAE version 2.0 grade will be analysed according to the grade present at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Maria De Santis, MD, Principal Investigator — Center for Oncology and Hematology Kaiser Franz Josef Hospital - Vienna - Austria; Stéphane Culine, MD, Principal Investigator — University Hospital St Louis - Paris - France
Locations (1):
- Pierre Fabre Research Institute, Boulogne, France

REFERENCES:
- [Derived] De Santis M, Wiechno PJ, Bellmunt J, Lucas C, Su WC, Albiges L, Lin CC, Senkus-Konefka E, Flechon A, Mourey L, Necchi A, Loidl WC, Retz MM, Vaissiere N, Culine S. Vinflunine-gemcitabine versus vinflunine-carboplatin as first-line chemotherapy in cisplatin-unfit patients with advanced urothelial carcinoma: results of an international randomized phase II trial (JASINT1). Ann Oncol. 2016 Mar;27(3):449-54. doi: 10.1093/annonc/mdv609. Epub 2015 Dec 16. PMID 26673352